CLINICAL TRIAL: NCT07029243
Title: Physical Prehabilitation With and Without Creatine/Whey Protein Supplementation Effects on Frailty In Patients With Cirrhosis
Brief Title: Prehab and Creatine/Whey Supplementation in Frailty Among Patients With Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 25-44010
Record Dates: First submitted 2025-05-15; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis; Frailty; Sarcopenia
Keywords: cirrhosis; liver; muscle; creatine; whey protein; frailty
MeSH Terms: conditions — Fibrosis; Frailty; Sarcopenia | interventions — Exercise; Nutritional Status; Creatine; Whey

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEAL-ME and placebo supplementation (Placebo Comparator): Patients within this arm will be administered the HEAL-ME digital app and placebo supplementation daily
  Interventions: Behavioral: HEAL-ME digital app; Dietary Supplement: Placebo
- HEAL-ME and creatine/whey protein supplementation (Experimental): Patients within this arm will be administered the HEAL-ME digital app and whey protein/creatine combination supplementation daily
  Interventions: Behavioral: HEAL-ME digital app; Dietary Supplement: Creatine supplementation; Dietary Supplement: Whey protein supplementation

INTERVENTIONS:
Behavioral: HEAL-ME digital app — HEAL-ME is a digital prehabilitation app that provides semi-guided nutrition/exercise prehabilitation
  Other Names: exercise; nutrition
Dietary Supplement: Creatine supplementation — Patients will take 5g creatine supplementation daily for 13 weeks
  Other Names: Creatine
  Arms: HEAL-ME and creatine/whey protein supplementation
Dietary Supplement: Whey protein supplementation — Patients will take 35g whey protein supplementation daily
  Other Names: Whey
  Arms: HEAL-ME and creatine/whey protein supplementation
Dietary Supplement: Placebo — Patients will be administered daily placebo supplementation.
  Arms: HEAL-ME and placebo supplementation

SUMMARY:
Frailty and muscle health are important for patients with chronic liver disease. This study looks at the use of a digital prehabilitation app (HEAL-ME) plus creatine and whey protein combination supplementation on maintaining muscle health in patients with liver disease. The investigators anticipate that this combination of supplementation and nutrition/exercise prehabilitation app will maintain muscle health in patients with liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cirrhosis by ICD-10 code, liver biopsy, abdominal imaging, or transient elastography
* Access to digital device and internet at home
* Ability to provide written informed consent before any study-related activities
* Ability to remain in study for at least 3 months

Exclusion Criteria:

* Allergy to milk protein
* On hemodialysis
* No English language proficiency
* Presence of condition or abnormality that in opinion of the Investigator will compromise safety of the patient or quality of the data
* Concomitant severe underlying systemic illness that in the opinion of the Investigator would interfere with completion of study
* Pregnant, breastfeeding, or intention of becoming pregnant during study time frame

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frailty | From enrollment to end of study at 12 weeks
  Frailty will be used to assess muscle quality. The liver frailty index (LFI) includes the measurement of grip strength, chair stands, and balance. The Liver Fraity Index typically ranges from 1.0 to 5.0 with the following cut-offs: Robust is Liver Frailty Index <3.2, Pre-frail is Liver Frailty Index between 3.2 and 4.4, and Frail is Liver frailty Index ≥4.4. We will use the previously identified cut-off of ≥4.4 (frail) vs. <4.4 (not frail) to identify frailty in this study.

SECONDARY OUTCOMES:
Feasibility: Completion Rate | From study enrollment to end of study at 12 weeks
  Completion rate will be assessed by study coordinators. Study coordinators will identify patients who do or do not complete the study during check-ins. Reasons for dropping out of the study will be recorded by study coordinators.
Health-related quality of life (HRQOL) | From enrollment to end of study at 12 weeks
  The Patient Reported Outcomes Measurement Information System (PROMIS)-29 v 2.0 is a NIH-supported effort to develop and disseminate patient-reported measures of HRQOL that has built-in normative reference to the US general population. The PROMIS-29 v2.0 will be used to assess HRQOL. A score ≤25 has been used to define the 25th percentile value for the general population and has previously been used in our studies to be considered poor HRQOL.
Self-Reported Physical Activity | From enrollment to end of study at 12 weeks
  The Duke Activity Status Index (DASI) will be used to measure self-reported physical activity. The DASI questionnaire provides a score from 0 to 58.2 with higher scores indicating better functional status and lower score indicating worse functional status. DASI will be measured as a continuous variable
Sarcopenia | From enrollment to end of study at 12 weeks
  Sarcopenia will be measured by abdominal computed tomography (CT) scan measured CT-quantified skeletal muscle index (skeletal muscle index (SMI) <50 cm2/m2 for men and <39 cm2/m2 for women). We have previously demonstrated that CT-quantified sarcopenia is associated with worse outcomes in patients with cirrhosis.
Feasibility: Adherence Rate | From study enrollment to end of study at 12 weeks
  Adherence rate will be assessed by study coordinators at each check-in. Adherence rate will include total adherence to the study protocol, adherence to supplement/placebo, and adherence to HEAL-ME activities.
Feasibility: Patient Satisfaction | From study enrollment to end of study at 12 weeks
  Patient satisfaction will be assessed by study coordinators at the end of the study. Patient satisfaction will be reported as a scalar variable from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lai, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No